CLINICAL TRIAL: NCT03004716
Title: Telemonitoring in Pulmonary Rehabilitation: Validity of a Remote Pulse Oxymetry System
Acronym: TELE-REHAB
Status: Completed | Type: Observational
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Other Study IDs: TELE-REHAB
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Pulmonary Rehabilitation; Telemedicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Aerobic training — 5 consecutive patients with chronicle obstructive pulmonary disease are offered to participate in the protocol when they have reached 45 min of aerobic training during their pulmonary rehabilitation program.
  During 5 sessions of 45 min, they are monitored with an oximeter device (Nonin 3150) which records heart rate (HR) and oxygen transcutaneous saturation (SpO2). The device also communicates with a telemedicine medical gateway which sends these data to a remote telemedicine center. Data are then provided on a secured online platform and compared with data recorded on the device (Nonin 3150).

SUMMARY:
The purpose of this study is to assess the feasibility and the reliability of a telemonitoring system during pulmonary rehabilitation in patients with chronicle obstructive pulmonary disease.

The feasibility is assessed using the patient's satisfaction and it ease of use.

The reliability of the remote telemonitoring system is assessed comparing the local data (extracted from the monitoring device itself) and the data transmitted through the telemonitoring platform.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years ;
* Chronicle obstructive pulmonary disease stage II/III/IV (FEV1 < 80%) ;
* Referred for pulmonary rehabilitation.

Exclusion Criteria:

* Pregnant woman or likely to be ;
* Patient under guardianship ;
* Neuropathic disorder ;
* Contraindication to cardiopulmonary exercise testing or pulmonary rehabilitation ;
* Progressive cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronicle obstructive pulmonary disease reffered for pulmonary rehabilitation.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Reliability between the heart rate (HR) acquired directly with the oximeter (Nonin 3150) and HR provided by the telemedicine gateway during the 1st session of 45 of aerobic training. | HR is assessed during a session of 45min for a total time frame 1h maximum.
  5 sessions of 45min of aerobic training will be carried out on 5 separate days (with a minimum of 1 day of rest between sessions) for a total time frame of 2 months. Data will be collected at the end of every session. Final endpoint will be the reliability of the data through study completion (5 sessions of 45min).
Reliability between the heart rate (HR) acquired directly with the oximeter (Nonin 3150) and HR provided by the telemedicine gateway during the 2nd session of 45 of aerobic training. | HR is assessed during a session of 45min for a total time frame 1h maximum.
  5 sessions of 45min of aerobic training will be carried out on 5 separate days (with a minimum of 1 day of rest between sessions) for a total time frame of 2 months. Data will be collected at the end of every session. Final endpoint will be the reliability of the data through study completion (5 sessions of 45min).
Reliability between the heart rate (HR) acquired directly with the oximeter (Nonin 3150) and HR provided by the telemedicine gateway during the 3rd session of 45 of aerobic training. | HR is assessed during a session of 45min for a total time frame 1h maximum.
  5 sessions of 45min of aerobic training will be carried out on 5 separate days (with a minimum of 1 day of rest between sessions) for a total time frame of 2 months. Data will be collected at the end of every session. Final endpoint will be the reliability of the data through study completion (5 sessions of 45min).
Reliability between the heart rate (HR) acquired directly with the oximeter (Nonin 3150) and HR provided by the telemedicine gateway during the 4th session of 45 of aerobic training. | HR is assessed during a session of 45min for a total time frame 1h maximum.
  5 sessions of 45min of aerobic training will be carried out on 5 separate days (with a minimum of 1 day of rest between sessions) for a total time frame of 2 months. Data will be collected at the end of every session. Final endpoint will be the reliability of the data through study completion (5 sessions of 45min).
Reliability between the heart rate (HR) acquired directly with the oximeter (Nonin 3150) and HR provided by the telemedicine gateway during the 5th session of 45 of aerobic training. | HR is assessed during a session of 45min for a total time frame 1h maximum.
  5 sessions of 45min of aerobic training will be carried out on 5 separate days (with a minimum of 1 day of rest between sessions) for a total time frame of 2 months. Data will be collected at the end of every session. Final endpoint will be the reliability of the data through study completion (5 sessions of 45min).

SECONDARY OUTCOMES:
Reliability between the transcutaneous saturation (SpO2) acquired directly with the oximeter (Nonin 3150) and SpO2 provided by the telemedicine gateway. | HR is assessed during 5 training sessions of 45min for a total time frame of 2month.
  5 sessions of 45min of aerobic training will be carried out on 5 separate days (with a minimum of 1 day of rest between sessions) for a total time frame of 2 months. Data will be collected at the end of every session. Final endpoint will be the reliability of the data through study completion (5 sessions of 45min).
Reliability of the telemedicine gateway in providing data. | 5 sessions of 45min will be carried out for 5 patients for a total time frame of 4months. For every patient, sessions will be carried out on 5 separate days (with a minimum of 1 day of rest between sessions).
  Data will be collected at the end of every sessions. Final endpoint will be the reliability of the telemedicine Gateway in providing data through study completion (5sessions of 45min for 5 different patients).
  Calculation : number of sessions provided by telemedicine gateway/number of scheduled sessions (n=25)
Patient's satisfaction assessed by Likert scale. | 5 sessions for 5 different patients will be assessed for a total time frame a 6month. Outcome will be assessed during the final session of every patient.
  Data will be presented as the patient's satisfaction of the system on the last of the 5 sessions at the end of the study.
Ability of the patients to be autonomous when using the device. | 5 sessions for 5 different patients will be assessed for a total time frame a 6month. Data will be collected after every sessions and presented as the number of patients autonomous when using the device.
  Number of patients autonomous when using the device will be presented for the the 2nd, 3rd, 4th and 5th session.

CONTACTS AND LOCATIONS:
Locations (1):
- ADIR Association, Bois-Guillaume, France

REFERENCES:
- [Derived] Bonnevie T, Gravier FE, Elkins M, Dupuis J, Prieur G, Combret Y, Viacroze C, Debeaumont D, Robleda-Quesada A, Quieffin J, Lamia B, Patout M, Cuvelier A, Muir JF, Medrinal C, Tardif C. People undertaking pulmonary rehabilitation are willing and able to provide accurate data via a remote pulse oximetry system: a multicentre observational study. J Physiother. 2019 Jan;65(1):28-36. doi: 10.1016/j.jphys.2018.11.002. Epub 2018 Dec 17. PMID 30573441